CLINICAL TRIAL: NCT00780767
Title: Angiojet Rheolytic Thrombectomy In Case of Massive Pulmonary Embolism A Prospective Single Center Feasibility and Safety Pilot Trial
Brief Title: Angiojet Rheolytic Thrombectomy in Case of Massive Pulmonary Embolism
Acronym: ART-MPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Robert F Bonvini, MD, University Hospital, Geneva
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Angiojet in MPE
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2008-10

CONDITIONS: Pulmonary Embolism
Keywords: angiojet; massive pulmonary embolism; RHEOLYTIC THROMBECTOMY; patients presenting with massive pulmonary embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thrombectomy arm (Experimental)
  Interventions: Device: ANGIOJET RHEOLYTIC THROMBECTOMY

INTERVENTIONS:
Device: ANGIOJET RHEOLYTIC THROMBECTOMY — The Angiojet catheter is a double lumen catheter percutaneously introduced via the common femoral vein into the main pulmonary trunk or the affected pulmonary artery respectively. One lumen serves to deliver high pressure saline jets into the thrombus and the other effluent lumen serves for clot removal utilizing a localized pressure region (Venturi effect) that attracts the thrombus for fragmentation into small particles. The fragmented debris are then pushed out through the evacuation line as a result of the retrograde high pressure saline jets, finally transporting them into a collection bag.

SUMMARY:
This pilot study is mainly aimed to evaluate the feasibility and safety of the percutaneous Angiojet Rheolytic Thrombectomy (ART) in patients presenting a MPE. Secondarily the effectiveness of this treatment modality will also be estimated.

DETAILED DESCRIPTION:
Pulmonary embolism (PE) is a major cause of mortality and morbidity in our society with more than 150.000 deaths every year in the US. Usually mortality occurs in the first hour after symptoms onset (up to 11%) and may further increase up to 17% at 3 months follow-up.

In case of massive PE (MPE) mortality dramatically increases up to 30% despite important improvements recently made in precocious diagnosis and aggressive medical treatments (i.e. i.v. thrombolysis).

Quite often (up to 40%) in case of PE there is at least one relative fibrinolysis contraindication, and less frequently these contraindications are absolute. In these quite rare cases, where thrombolytic therapy is absolutely contraindicated, a surgical thrombo-embolectomy is advised, however this kind of challenging surgery is not available world-wide and it still remains associated with a prohibitive high rate of mortality.

A less invasive alternative remains the percutaneous thrombectomy, which may further be divided into:

* Aspiration thrombectomy,
* Fragmentation thrombectomy,
* Rheloytic thrombectomy. The first transvenous percutaneous pulmonary embolectomy was performed more than 30 years ago; however, it is only recently that, thanks to new developed technologies, phyisicians manifest an increased interest in developing this promising less invasive procedure.

The angiojet rheolytic thrombectomy (ART) catheter (Angiojet : Possis medical ; Minneapolis, MN, USA) utilizes high velocity saline jets for thrombus aspiration, maceration and evacuation through the Bernoulli principle. Nowadays this technology is successfully utilized daily in the coronary and peripheral artery fields (i.e. thrombus aspiration during coronary or arterial angioplasty).

Due to its safety and efficacy, demonstrated in randomized trials including patients with coronary artery disease, several recent reports also confirmed the usefulness of this ART also in extra-coronary domain (peripheral arterial and venous diseases).

Massive PE, as the thrombotic coronary artery occlusion, is a life threatening clinical manifestation, therefore several centers began to manage it associating mechanical (i.e.ART) clot removal and pharmacological (i.e. lysis).

The first small, retrospective non randomized series suggest the safety and efficacy of this technology, confirming its feasibility compared with the actual proposed treatment of MPE (i.e. i.v. or in-situ pulmonary thrombolysis).

The first in man utilization of the Angiojet rheolytic thrombectomy for treating acute massive PE dates 1997, however in-vitro tests also revealed that Angiojet is able to successfully remove thrombus up to 14 days old, thus enlarging its usefulness also in sub-acute cases (i.e.>14 days old thrombus).

Despite the fact that indication of an i.v. fibrinolysis is worldwide accepted in case of MPE and that established lysis protocols are nowadays available, mortality remains unacceptably high (up to 30%) and bleeding related morbidity a major concern. In fact in large PE registries, up to 20% of the patients experienced major bleedings complications, and in 3% of the cases this was intracranial.

Of interest in case of sub-massive PE (sub-MPE), which is also associated with a quite high mortality (up to 8%) some disagreement concerning the best treatment modality still persists. Several authors support an intensive treatment modality favourizing the systemic i.v. thrombolysis; however, others suggest a more conservative attitude (anticoagulation alone with fibrinolysis only in case of clinical deterioration). These cases of sub-MPE may be very challenging, because an established consensus of the definition of sub-MPE combining clinical, radiological and cardiological criteria are still lacking. Furthermore the thrombolytic regimen is not complication-free, suggesting that, before performing an i.v. thrombolysis, the physician in charge of the patient has to seriously take in consideration all the absolute and the relative contra-indications of such a treatment. (i.e.recent surgery, active peptic ulcer, intra-cerebral bleeding, pregnancy, neoplasm, see Table 1).

The ongoing debate on how to improve mortality in patients with MPE and concerning the correct managing of patients with sub-MPE suggests that in both cases, there is an urgent need of improving the actual treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged >18 years old
2. Patients presenting a MPE (i.e. hemodynamically unstable at moment of the inclusion (i.e. shock index (SI) >1).
3. Patients where a hemodynamic stability (SI=1) is hardly obtained despite increasing dose of drug support.

   * If after 2 hours from the first medical contact where an intensive fluid substitution and cathecolamine support is begun the patient remains with a SI = 1, he/she could be included in the ART protocol.
   * If after an initial successful drug support (fluid + catecholamine) the patient represents a second episode of hemodynamic instability, he/she could be included in the ART protocol.
   * If the patient is under chronic negative chronotrope medication (e.g.beta-blockers) a SI = 1 will be sufficient to include the patient in the study
4. The MPE have to be confirmed by thorax CT-scan or suspected by echocardiography (i.e.visualized thrombus on the RV or main pulmonary trunk or RV overload with a high clinical suspicion of MPE).

Exclusion Criteria:

1. Very unstable patients with life threatening MPE where the time delays to transport them in the cathterization laboratory (i.e. <30 minutes) to perform the ART procedure is not acceptable because the systemic i.v. thrombolysis have to be immediately initiated in the emergency department.
2. Patients where a percutaneous right heart catheterization via the common femoral vein is contraindicated (e.g.vascular malformation, inferior cava vein occlusion, presence of bilateral ilio-femoral thrombosis, RV or pulmonary trunk malformation).
3. Patients with sub-MPE without any other clinical or para-clinical sign of severity (e.g. haemodynamically stable = SI<1).
4. Patients where the clinical evaluation estimated that the observed episode of MPE is older than 14 days (i.e. sub-acute phase with organized thrombus = ART less efficacious).
5. Patient with an estimated clearance to creatinine less than 30 ml/min.
6. Patients or members of their family who refused to give their signed informed consenstement.
7. Patient haemodynamically very unstable where the first clinical evaluation concludes that every therapeutic effort including the ART procedure or a systemic fibrinolysis will not change the short-term prognosis of the patient (i.e. imminent death).
8. Patients with a life expectancy of <3months for other medical pre-existing conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Successfully perform an ART in all patients presenting a MPE = technical feasibility of ART | 1 month
No major device-related complications, no major procedure-related complications = safety of ART | 1 month

SECONDARY OUTCOMES:
Improve the clinical, haemodynamic and the radiological issues of the treated patients | 1 month
Evaluate the clinical status, and the echocardiographic parameters at 3 months | 1 month
Analyze the technical aspect of the ART procedure | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Univesity hospital of geneva, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Result] Margheri M, Vittori G, Vecchio S, Chechi T, Falchetti E, Spaziani G, Giuliani G, Rovelli S, Consoli L, Biondi Zoccai GG. Early and long-term clinical results of AngioJet rheolytic thrombectomy in patients with acute pulmonary embolism. Am J Cardiol. 2008 Jan 15;101(2):252-8. doi: 10.1016/j.amjcard.2007.07.087. PMID 18178417
- [Derived] Bonvini RF, Roffi M, Bounameaux H, Noble S, Muller H, Keller PF, Jolliet P, Sarasin FP, Rutschmann OT, Bendjelid K, Righini M. AngioJet rheolytic thrombectomy in patients presenting with high-risk pulmonary embolism and cardiogenic shock: a feasibility pilot study. EuroIntervention. 2013 Apr 22;8(12):1419-27. doi: 10.4244/EIJV8I12A215. PMID 23680957